CLINICAL TRIAL: NCT06651463
Title: Evaluation of the Feasibility of Camera Measurement of Colorimetric Parameters of the Brain During Neurosurgery Operations: Tissue Oximetry and Endogenous or Induced Fluorescence
Acronym: NEUROVISION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL24_0709
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Brain Diseases
Keywords: feasibility; tissue identification; neurosurgery; video
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video Capture (Experimental): Brain of patients, presenting a brain pathology eligible for a neurosurgery operation requiring a standard functional and/or histological diagnosis at HCL, will be video recorded with colorimetric cameras in order to evaluate the feasibility of identifying tissue.
  Interventions: Other: Videorecording

INTERVENTIONS:
Other: Videorecording — Two cameras will be used to make the recordings: a classic camera placed on a stand 1 meter from your head, outside the sterile area and the color camera of the microscope used for the surgery.

SUMMARY:
The management of many brain pathologies involves obtaining a functional and histological diagnosis and performing neurosurgery when possible. Histological diagnosis makes it possible to differentiate healthy areas from pathological areas. Functional diagnosis allows the identification of brain areas to be spared during neurosurgery in order to avoid any permanent post-operative disability.

The visual analysis of the color and texture of the brain by the trained eye of the neurosurgeon is largely part of his operating practice. It allows it to differentiate between healthy and pathological areas. Likewise, color variations linked to the functional activation of brain areas are sometimes visible to the naked eye. However, this approach is not optimal due to the limits of human vision. It is also very strongly dependent on the experience and expertise acquired by the neurosurgeon. This approach is therefore largely limited in many operating contexts: low visual contrasts, less experienced neurosurgeon.

ELIGIBILITY:
Inclusion Criteria:

* Adult from both sex
* Neurosurgery requiring a functional diagnosis by cortical electrical stimulation OR a histological diagnosis with or without fluorescent agent (5-ALA) for a tumor pathology or epilepsy or an arteriovenous malformation.
* Patient able to sign a non-opposition

Exclusion Criteria:

* Impaired renal function defined by the presence of creatinine clearance less than 30ml/min
* Patient under treatment with beta-blocker
* Contraindication to performing an MRI (pacemaker)
* Contraindication to the use of electrical cortical stimulation
* History of life-threatening allergic reactions or known hypersensitivity to 5-ALA
* Pregnant, breastfeeding woman
* Subject participating in another interventional research including an exclusion period still ongoing at pre-inclusion,…
* Persons deprived of liberty by a judicial or administrative decision
* People receiving psychiatric care
* Persons admitted to a health or social establishment for purposes other than research
* Adults subject to a legal protection measure (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recording video of useful quality to determine tissue quality | Video will be recodered during surgery and feasibility will be assessed once all the video of all included patients will be recorded. 2-3 hours
  The technical feasibility of the measurement will be determined by obtaining videos of sufficient quality to reach the detection threshold of the various functional and pathological markers. We will test the technical feasibility based on the expertise of the operator (researcher from the scientific team or operating room staff). This quality of the data will be judged using the expertise of CREATIS researchers. This quality is based on criteria linked to contrasts, signal-to-noise ratios, the absence of specular reflection artifacts and image movement. The evaluation methods which will be used during the meetings will be inspired by standard approaches from our previous work in collaboration with HCL

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pierre Wertheimer, Bron, France